CLINICAL TRIAL: NCT07254546
Title: GRAtitude et Considération Envers Les Donneurs Vivants du Rein
Brief Title: A Qualitative Study on Gratitude and Recognition Toward Living Kidney Donors
Acronym: GRACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP251133
Record Dates: First submitted 2025-11-18; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Kidney Transplantation; Nephrectomy,Kidney Donation
Keywords: Incentive; Living donor; Living donor nephrectomy; Living kidney donation; Gratitude

STUDY DESIGN:
Intervention Model Description: Monocentric cohort of Living donors of Kidney
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Living donors of Kidney (Other): This cohort includes individuals who have donated a kidney at Hôpital Saint-Louis between January 1, 2020, and December 31, 2025, as well as individuals currently engaged in a living kidney donation process with a nephrectomy planned before June 30, 2026, in the same institution. Participants will take part in semi-structured qualitative interviews exploring their perceptions and experiences related to post-donation recognition.
  Interventions: Behavioral: Semi-structured qualitative interview

INTERVENTIONS:
Behavioral: Semi-structured qualitative interview — Participants will take part in a one-on-one semi-structured qualitative interview exploring their experiences and perceptions related to living kidney donation and potential forms of post-donation recognition.
  The interview guide includes open-ended questions addressing:
  * Personal motivations for donation;
  * Emotional and relational experiences throughout the donation process;
  * Ethical perceptions of living donation;
  * Views on symbolic recognition (e.g., commemorative medal, public acknowledgment, ceremony);
  * Perceptions of paired kidney donation (KPD);
  * Social representations of living donation in their personal environment and in society.
  Interviews will last approximately 45 to 60 minutes and will be conducted either in person at Hôpital Saint-Louis or via secure videoconference.
  All interviews will be recorded, transcribed verbatim, anonymized, and analyzed using inductive thematic analysis (NVivo or equivalent software).

SUMMARY:
Kidney transplantation is widely recognized as the best treatment for patients with end-stage renal disease. However, its development is limited by the persistent shortage of available organs. Living donor kidney transplantation offers the best functional and survival outcomes, yet the number of procedures remains insufficient.

Living kidney donation relies on a voluntary and altruistic act by a healthy individual who accepts surgery without direct medical benefit. This act of generosity raises important questions regarding how society acknowledges and values such commitment. The lack of formal recognition may contribute to the psychological burden experienced by some donors and may not adequately reflect the gratitude of the medical community and society toward them.

This study aims to explore the perceptions of living kidney donors regarding the potential implementation of a symbolic form of recognition (for instance, a commemorative medal) offered after donation. The hypothesis is that such recognition could improve donors' post-donation experience and strengthen the societal value associated with living organ donation, while fully respecting ethical principles prohibiting any financial reward.

This is a qualitative, monocentric study based on semi-structured interviews with individuals who have donated a kidney. The interviews will focus on donors' motivations, their personal experience of donation, and their opinions about different possible forms of post-donation recognition. Interviews will be recorded, transcribed verbatim, and analyzed using inductive thematic analysis to identify recurring themes and perspectives.

The main endpoint is the identification of thematic categories related to donors' perception of post-donation recognition and its potential impact on their experience. Secondary objectives include exploring donors' expectations regarding societal gratitude, their views on the symbolic value of such recognition, and the potential influence on future donor engagement.

The findings of this study are expected to contribute to the ethical reflection surrounding the acknowledgment of living donors, support initiatives promoting non-financial recognition, and help develop respectful and meaningful ways of expressing societal gratitude toward those who make the gift of life possible.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have donated a kidney at Hôpital Saint-Louis between January 1, 2020, and December 31, 2025, or are currently engaged in a living kidney donation process with nephrectomy scheduled before June 30, 2026.
* Age ≥ 18 years.
* Able to provide informed consent.

Exclusion Criteria:

* Refusal or opposition to participate in the study.
* Individuals under legal protection (guardianship, curatorship, or legal safeguard).
* Individuals deprived of liberty by judicial or administrative decision.
* Individuals under 18 years of age.
* Kidney donation performed in a hospital other than Hôpital Saint-Louis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Themes related to donor perceptions of post-donation recognition | At baseline
  Inductive thematic analysis of semi-structured interviews with living kidney donors, identifying key themes and subthemes related to their perception of post-donation recognition or symbolic rewards (e.g., commemorative medal, public acknowledgment).

SECONDARY OUTCOMES:
Perceptions of Kidney Paired Donation (KPD) | At baseline
  Exploration of participants' views and emotional responses toward kidney paired donation programs, including ethical and logistical aspects.
  A semi-structured interview lasting 30-60 minutes, either in person during another scheduled treatment or via videoconference.
Initial Motivations for Donation | At baseline
  Identification of personal, relational, or altruistic motivations that led participants to consider or complete living kidney donation.
  A semi-structured interview lasting 30-60 minutes, either in person during another scheduled treatment or via videoconference.
Experience of the Donation Pathway | At baseline
  Evaluation of participants' experiences throughout the donation process, including emotional journey, perceived support, and acknowledgment by healthcare professionals.
  A semi-structured interview lasting 30-60 minutes, either in person during another scheduled treatment or via videoconference.
Ethical Perceptions of Living Donation and Symbolic Recognition | At baseline
  Analysis of ethical reflections expressed by donors regarding the concept of recognition, symbolic rewards, or institutional gratitude (e.g., medals, diplomas, ceremonies).
  A semi-structured interview lasting 30-60 minutes, either in person during another scheduled treatment or via videoconference.
Social Representations of Living Donation | At baseline
  Investigation of how donors perceive societal and familial views about living kidney donation, including stigma, admiration, or misunderstanding.
  A semi-structured interview lasting 30-60 minutes, either in person during another scheduled treatment or via videoconference.
Barriers or Reluctance Toward Kidney Paired Donation | At baseline
  Identification of logistical, emotional, or ethical barriers expressed by participants regarding paired exchange donation.
  A semi-structured interview lasting 30-60 minutes, either in person during another scheduled treatment or via videoconference.

IPD SHARING:
Plan to Share IPD: Undecided